CLINICAL TRIAL: NCT02456545
Title: Improving Early Recognition and Intervention in At-risk Stages of Bipolar Disorders
Acronym: BipoLife-A1
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Charite University, Berlin, Germany (Other); Ruhr University of Bochum (Other); Goethe University (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Philipps University Marburg (Other); University Hospital Tuebingen (Other); Vivantes Hospital am Urban, Berlin (Unknown)
Responsible Party: Principal Investigator, Andrea Pfennig, Prof. Dr. med. Andrea Pfennig, Technische Universität Dresden
Other Study IDs: BipoLife-A1
Record Dates: First submitted 2015-05-11; First posted 2015-05-28 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- help-seekers at-risk: persons consulting collaborating Early Recognition Centers presenting with hints for ≥ 1 potential risk factor for BD (e.g. (sub)threshold affective symptomatology, anxiety, sleep disturbances, family history, episodic substance misuse, ADHD)
  anticipated n = 500
  Interventions: Other: ≥ 1 potential risk factor for BD
- patients with depressive syndrome: in- and outpatients with depressive syndrome (SCID)
  anticipated n = 500
  Interventions: Other: depressive syndrome
- patients with ADHD: in- and outpatients with Attention-Deficit/Hyperactivity-Disorder (ADHD)
  anticipated n = 150
  Interventions: Other: ADHD
- representative population cohort: representative population cohort from the IMAGEN study
  anticipated n = 500

INTERVENTIONS:
Other: ≥ 1 potential risk factor for BD — exposure to ≥ 1 potential risk factors for BD (e.g. (sub)threshold affective symptomatology, anxiety, sleep disturbances, family history, episodic substance misuse)
  Groups: help-seekers at-risk
Other: depressive syndrome — in- and outpatients with depressive syndrome
  Groups: patients with depressive syndrome
Other: ADHD — in- and outpatients with ADHD
  Groups: patients with ADHD

SUMMARY:
Prospective multicentre observational study for treatment approaches in at-risk individuals. Furthermore the purpose of this study is to test feasibility of a clinical staging model and validate diagnostic tools to identify individuals at risk state for the development of BD.

DETAILED DESCRIPTION:
This project is one out of nine projects and four translational platforms forming the core of an interdisciplinary consortium to research on the most important areas of uncertainties and unmet needs in early recognition and diagnostic assessment, prevention of relapse, and therapeutic strategies of BD.

Within this project, currently used diagnostic tools for subthreshold bipolar symptoms (BPSS-P, EPIbipolar, BAR criteria) will be deployed within the first 24 months in defined risk groups. Predictive power of individual risk factors/risk constellations will be determined regarding the manifestation and prodromal development of BD within ≥24 months (follow-up every 6 months). Potential resilience factors are ascertained. Additionally, the diagnostic tools will be used in a representative cohort (IMAGEN, to ascertain the prevalence of clinical/neurobiological at-risk constellations in non-selected youth and young adults, data from previous follow-ups will be used, suffering/help-seeking behavior will be assessed). Regarding treatment, at-risk subjects identified will be staged according to a pilot staging model. Treatment guidance is provided linked to the model, however, the naturalistic setting allows for individual decision making. Reasons for decisions will be ascertained, efficacy will be assessed with respect to symptomatology, psychosocial functioning and conversion to full BD, tolerability/safety will be assessed according to research standard. Outcomes will be assessed within ≥ 24 months. Using the results, the clinical staging model & guidance will be refined. The long-term goal is to provide a model for research and clinical initiatives.

Synopsis of study goals:

1. Determination of the predictive power of individual risk factors and risk constellations in defined risk groups for BD,
2. Identification of resilience factors,
3. Integration of results for further development of diagnostic tools and harmonization of the diagnostic process across centers,
4. Investigation of the process of treatment decision making, efficacy (acute/preventive effects) and tolerability/safety in at-risk subjects in a naturalistic setting, testing the feasibility of a pilot clinical staging model with treatment guidance,
5. Refinement of the staging model and guidance.

ELIGIBILITY:
Inclusion Criteria:

* Risk group I: help-seeking persons consulting collaborating Early Recognition Centers presenting hints for ≥ 1 potential risk factor for BD (e.g. (sub)threshold affective symptomatology, anxiety, sleep disturbances, family history of bipolar disorder, episodic substance misuse, depressive syndrome)
* Risk group II: in- and outpatients with depressive syndrome (SCID) from the network sites
* Risk group III: in- and outpatients with ADHD already cared for in the Dept. of Child and Adolescent as well as Adult psychiatry in Würzburg
* Representative population cohort: IMAGEN study participants

Exclusion Criteria:

* bipolar disorder
* schizaffective disorder
* schizophrenia
* dominating anxiety disorder, obsessive-compulsive disorder
* dominating substance-related disorder

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Risk groups I: help-seeking persons with subthreshold symptoms
  Risk group II: in- and outpatients with depressive disorder
  Risk group III: in- and outpatients with ADHD
  representative population cohort from IMAGEN study
Sampling Method: Non-Probability Sample
Enrollment: 1419 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Prodromal Symptoms for bipolar development via BPSS-FP & EPIbipolar | baseline
  * Bipolar Prodrome Symptom Scale - Full Prospective - BPSS-FP describes and rates prodromal mania/depression and other symptoms that have occurred in the past month and in the past year;
  * Early Phase Inventory for bipolar disorders - EPIbipolar describes and rates symptoms associated with BD in the early phase (past 12 months) as sleep and circadian rhythm, mood swings and neuroticism, anxiety, functioning and comorbidity in childhood and youth, substance use, development of symptomatic pattern
Prodromal Symptoms for bipolar development via BPSS-FP & EPIbipolar | 1-year follow-up
  * Bipolar Prodrome Symptom Scale - Full Prospective - BPSS-FP describes and rates prodromal mania/depression and other symptoms that have occurred in the past month and in the past year;
  * Early Phase Inventory for bipolar disorders - EPIbipolar describes and rates symptoms associated with BD in the early phase (past 12 months) as sleep and circadian rhythm, mood swings and neuroticism, anxiety, functioning and comorbidity in childhood and youth, substance use, development of symptomatic pattern
Prodromal Symptoms for bipolar development via BPSS-FP & EPIbipolar | 2-year follow-up
  * Bipolar Prodrome Symptom Scale - Full Prospective - BPSS-FP describes and rates prodromal mania/depression and other symptoms that have occurred in the past month and in the past year;
  * Early Phase Inventory for bipolar disorders - EPIbipolar describes and rates symptoms associated with BD in the early phase (past 12 months) as sleep and circadian rhythm, mood swings and neuroticism, anxiety, functioning and comorbidity in childhood and youth, substance use, development of symptomatic pattern
Diagnostic Status: psychiatric disorders via SCID-I | baseline
  Diagnostic Status: psychiatric disorders via SCID-I
Diagnostic Status: psychiatric disorders via SCID-I | 1-year follow-up
  Diagnostic Status: psychiatric disorders via SCID-I
Diagnostic Status: psychiatric disorders via SCID-I | 2-year follow-up
  Diagnostic Status: psychiatric disorders via SCID-I

SECONDARY OUTCOMES:
Psychotic Prodrome via PQ-16 (SOPS, SPi-A) | baseline
  Screening for psychotic prodrome using Prodromal Questionnaire - PQ-16
  Assessing psychotic prodrome after positive screening via Structured Interview for Prodromal Syndroms - SOPS and Schizophrenia Proneness Instrument, Adult Version - SPi-A (german version)
Personality disorder via SCID-II (screening) | baseline
  self-report screening questionnaire for personality disorder via SCID-II
  Assessing personality disorder via SCID-II after positive screening
Depressive Symptoms via Montgomery-Åsberg Depression Rating Scale (MADRS) | baseline
  Clinician-rated severity of depressive symptoms over the past 7 days, 10 items, scoring 0-6 each, yielding a total between 0 and 60.
Depressive Symptoms via Quick Inventory of Depressive Symptomatology (QIDS-SR16) | baseline
  Self-rated severity of depressive symptoms over the past 7 days, 16 items, scoring 0-3 each, yielding a total between 0 and 48.
Manic Symptoms via Young Mania Rating Scale (YMRS) | baseline
  Clinician-rated severity of manic symptoms over the past 48 hours, 11 items, 7 items scoring 0-4 each,4 items scoring 0-8 each, yielding a total between 0 and 60.
Manic Symptoms via Altman Self-Rating Mania Scale (ASRM) | baseline
  Self-rated severity of manic symptoms over the past 7 days, 5 items, scoring 0-4 each (0=no difficulty, 3=severe difficulty), yielding a total between 0 and 50.
Functional Impairment via Functioning Assessment Short Test (FAST) | baseline
  Clinician-rated functional impairment over the past 48 hours, 24 items, scoring 0-3 each (0=no difficulty, 3=severe difficulty), yielding a total between 0 and 72.
Functional Impairment via Functioning Assessment Short Test (FAST) | 1-year follow-up
  Clinician-rated functional impairment over the past 48 hours, 24 items, scoring 0-3 each (0=no difficulty, 3=severe difficulty), yielding a total between 0 and 72.
Functional Impairment via Functioning Assessment Short Test (FAST) | 2-year follow-up
  Clinician-rated functional impairment over the past 48 hours, 24 items, scoring 0-3 each (0=no difficulty, 3=severe difficulty), yielding a total between 0 and 72.
Functioning via GAF-scale | baseline
  Clinician-rated global functioning at the present moment via Global Assessment of Functioning scale (GAF-scale), scoring between 1-100 (1=no difficulty, 100=Persistent danger of severely hurting self or others or persistent inability to maintain minimal personal hygiene or serious suicidal act with clear expectation of death)
Functioning via GAF-scale | 1-year follow-up
  Clinician-rated global functioning at the present moment via Global Assessment of Functioning scale (GAF-scale), scoring between 1-100 (1=no difficulty, 100=Persistent danger of severely hurting self or others or persistent inability to maintain minimal personal hygiene or serious suicidal act with clear expectation of death)
Functioning via GAF-scale | 2-year follow-up
  Clinician-rated global functioning at the present moment via Global Assessment of Functioning scale (GAF-scale), scoring between 1-100 (1=no difficulty, 100=Persistent danger of severely hurting self or others or persistent inability to maintain minimal personal hygiene or serious suicidal act with clear expectation of death)
Impulsiveness via Barrat Impulsiveness Scale (BIS) | baseline
  Self-rated measure of impulsiveness, 30 items, scoring 1-4 each (1=rarely/never, 4=almost always/always), yielding a total between 30 and 120.
Traumatic life events in childhood via Childhood Trauma Questionnaire (CTQ-SF) | baseline
  Retrospective self-report to identify adolescent and adult clients with histories of trauma, 28 items, scoring on a 5-point Likert-type scale according to the frequency with which experiences occurred ("never true" to "very often true").
Affective temperament via Temperament Evaluation of Memphis, Pisa, Paris, and San Diego-Autoquestionnaire version (TEMPS-A) | baseline
  Self-rated assessment of five affective temperaments, 30 items, dichotomous scale 0="applies", 1= "does not apply".
Creativity via Barron Welsh Art Scale (BWAS) | baseline
  Assessment of the aesthetic preference by scoring "like" or "dislike" for certain black-and-white figures (85 items).
Creative Achievement via Creative Achievement Questionnaire (CAQ) | baseline
  Self-report measure of creative achievements across 10 domains, 96 items.
Chronic Stress via Trierer Inventar zum chronischen Stress (TICS) | baseline
  Self-rated measure of chronic stress in the past 3 months, 57 items, scoring 0-4 each (1=never, 4=almost always), yielding a total between 0 and 228.
Ressources and self-management via Fragebogen zur Erfassung von Ressourcen und Selbstmanagementfähigkeit (FERUS) | baseline
  Self-rated measure of health related ressources and self-management ability in the past two to three weeks, 66 items, scoring 1-5 each (1=strongly disagree, 4=strongly agree), yielding a total between 66 and 330.
Quality of life via WHOQOL-BREF | baseline
  Self-rated measure to assess subjective quality of life in the past two weeks, 26 items, 5-point scale with varying verbal equivalents
Quality of life via WHOQOL-BREF | 1-year follow-up
  Self-rated measure to assess subjective quality of life in the past two weeks, 26 items, 5-point scale with varying verbal equivalents
Quality of life via WHOQOL-BREF | 2-year follow-up
  Self-rated measure to assess subjective quality of life in the past two weeks, 26 items, 5-point scale with varying verbal equivalents
Sensitivity of Behavioral Inhibition System and Behavioral Activation System via BIS/BAS scales | baseline
  Self-rated measure to assess Sensitivity of the Behavioral Inhibition System and the Behavioral Activation System, 24 items, scoring 1-4 each (1=strongly disagree, 4=strongly agree) yielding a total between 24 and 96.
Life events and -changes via Life Events Questionnaire (LEQ) | baseline
  Inventory to assess life events and -changes during the past year, 82 items, choosing applying life events from a list of 82 events, rating Type of effect (good vs bad) and effect of event on life (0=no effect, 3=great effect).
Life events and -changes via Life Events Questionnaire (LEQ) | 1-year follow-up
  Inventory to assess life events and -changes during the past year, 82 items, choosing applying life events from a list of 82 events, rating Type of effect (good vs bad) and effect of event on life (0=no effect, 3=great effect).
Life events and -changes via Life Events Questionnaire (LEQ) | 2-year follow-up
  Inventory to assess life events and -changes during the past year, 82 items, choosing applying life events from a list of 82 events, rating Type of effect (good vs bad) and effect of event on life (0=no effect, 3=great effect).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pfennig, Dr. med., Principal Investigator — University Hospital Dresden, Technische Universität Dresden; Michael Bauer, Dr. rer. nat., Principal Investigator — University Hospital Dresden, Technische Universität Dresden; Martin Lambert, Dr. med., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (9):
- Germany (9):
  - Charite University Berlin, Berlin
  - Vivantes Hospital am Urban, Berlin
  - Ruhr University of Bochum, Bochum
  - University Hospital Dresden, Präventionsambulanz mit Früherkennungszentrum, Dresden
  - University Hospital Frankfurt, Frankfurt a.M.
  - University Hospital Hamburg-Eppendorf, Hamburg
  - Philipps University of Marburg Medical Center, Marburg
  - Ruppiner Kliniken, Klinik für Psychiatrie, Psychotherapie und Psychosomatik, Neuruppin
  - University Hospital Tuebingen, Tübingen

REFERENCES:
- [Background] Bechdolf A, Ratheesh A, Wood SJ, Tecic T, Conus P, Nelson B, Cotton SM, Chanen AM, Amminger GP, Ruhrmann S, Schultze-Lutter F, Klosterkotter J, Fusar Poli P, Yung AR, Berk M, McGorry PD. Rationale and first results of developing at-risk (prodromal) criteria for bipolar disorder. Curr Pharm Des. 2012;18(4):358-75. doi: 10.2174/138161212799316226. PMID 22239567
- [Background] Correll CU, Olvet DM, Auther AM, Hauser M, Kishimoto T, Carrion RE, Snyder S, Cornblatt BA. The Bipolar Prodrome Symptom Interview and Scale-Prospective (BPSS-P): description and validation in a psychiatric sample and healthy controls. Bipolar Disord. 2014 Aug;16(5):505-22. doi: 10.1111/bdi.12209. Epub 2014 May 8. PMID 24807784
- [Background] Leopold K, Ritter P, Correll CU, Marx C, Ozgurdal S, Juckel G, Bauer M, Pfennig A. Risk constellations prior to the development of bipolar disorders: rationale of a new risk assessment tool. J Affect Disord. 2012 Feb;136(3):1000-10. doi: 10.1016/j.jad.2011.06.043. Epub 2011 Jul 30. PMID 21802741
- See also: further patient information — https://www.bipolife.org/
- See also: Project providing participants from representational cohort — http://www.imagen-europe.com/